CLINICAL TRIAL: NCT06661018
Title: The Effect of Coenzyme Q10 Supplementation on Global Longitudinal Strain Values in Acute ST Segment Elevation Myocardial Infarction Patients Treated With Primary Percutaneous Coronary Intervention
Brief Title: Effect Supplementation of COenzyme Q10 in Acute STEMI Underwent PPCI
Acronym: ESCOMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Ilham Uddin, MD, Principal Investigator, Universitas Diponegoro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1648/EC/KEPK-RSDK/2023
Record Dates: First submitted 2024-10-17; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: ST Segment Elevation Myocardial Infarction (STEMI); Coenzyme Q10
Keywords: coenzyme Q10; Acute Myocardial Infarction; ST Segment Elevation Myocardial Infarction (STEMI); Global Longitudinal Strain; Ubiquinone; Primary Percutaneous Coronary intervention; Cardiovascular disease
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Cardiovascular Diseases | interventions — coenzyme Q10; Ubiquinone

STUDY DESIGN:
Intervention Model Description: This research is an experimental clinical study with a double blinded randomized controlled trial design. The study group consisted of patients with acute STEMI underwent primary PCI. The first group was patients who received standard treatment plus coenzyme Q10 100mg / 12 hours orally for up to 8 weeks (group A). Meanwhile, the second group was patients who received standard treatment plus placebo for up to 8 weeks (group B).
Who Masked: Participant, Care Provider, Investigator
Masking Description: participant, care Provider, and investigator will not know either they include in treatment or control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Oral Coenzyme Q10) (Experimental): Experimental: Group A (Oral Coenzyme Q10) Participants who received standard treatment plus Coenzyme Q10 100 mg / 12 hours orally for up to 8 weeks.
  Intervention/Treatment Drug: Oral Coenzyme Q10
  * Participants will be randomized into group receiving either oral Coenzyme Q10 or placebo for up to 8 weeks
  Interventions: Drug: Coenzyme Q 10
- Group B (Placebo) (Placebo Comparator): Placebo Comparator: Group B (Placebo) Participants who received standard treatment plus Placebo / 12 hours orally for up to 8 weeks.
  Intervention/Treatment Drug: Placebo
  * Participants will be randomized into group receiving either oral Coenzyme Q10 or placebo for up to 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Coenzyme Q 10 — participant will receive STEMI standard treatment plus oral Coenzyme Q10 (chewable tablet) 100 mg / 12 hours for 8 weeks
  Other Names: CoQ10; ubiquinone
  Arms: Group A (Oral Coenzyme Q10)
Drug: Placebo — participant will receive STEMI standard treatment plus placebo /12 hours for 8 weeks
  Arms: Group B (Placebo)

SUMMARY:
Left ventricular remodeling can still occur after primary percutaneous coronary intervention (PCI). Global longitudinal strain (GLS) assessment has been used as a predictor of left ventricular remodeling. Coenzyme Q10 is known for its anti-inflammatory and antioxidant properties, which may help reduce cardiac remodeling. This study aims to determine the effect of CoQ10 administration after myocardial infarction as an adjunct to standard therapy on left ventricular remodeling, assessed through changes in GLS values.

Researchers will compare Coenzyme Q10 to a placebo to see if Coenzyme Q10 has a greater effect on improving left ventricular GLS values in patients with ST-Elevation Myocardial Infarction undergoing primary percutaneous coronary intervention.

DETAILED DESCRIPTION:
This is a randomized, double blind study with 2 treatment groups. Participants diagnosed with Acute STEMI post primary PCI who meet the inclusion criteria and no exclusion criteria are given an explanation regarding the research and additional therapy that will be given, then informed consent is requested. Participants will be randomized to one of the two treatment groups by chance. Patients randomized to the first group will receive coenzyme Q10 100mg/12hours. Patients randomized to the other treatment group will receive a placebo. It is expected that the patients of the treatment group with the coenzyme Q10 will have a greater improvement of their GLS.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 - 80 years
* Agree to participate in the study
* Patients with a diagnosis of Acute Myocardial Infarction with ST-Segment Elevation (AMI-STE) with onset < 12 hours who underwent primary percutaneous coronary intervention (PCI)
* Successful primary PCI on the culprit lesion (residual stenosis < 20%, TIMI flow III)
* Received standard medication therapy according to guidelines (Guideline-Directed Medical Therapy; GDMT) achieved during hospitalization
* Sinus rhythm at the time of echocardiographic examination

Exclusion Criteria:

* Patients who routinely consume CoQ10 prior to the study
* Patients with hemodynamic conditions of Killip class III-IV and NYHA class III-IV
* Patients with a history of previous acute myocardial infarction
* Patients with a history of previous PCI or fibrinolytic therapy
* Patients with a history of previous coronary artery bypass surgery
* Patients with heart valve disease greater than moderate severity
* Patients receiving warfarin therapy
* Patients with a diagnosis of isolated right ventricular infarction
* Patients with inadequate echocardiographic image quality (poor echo window)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male and female gender that aligns with the sex they were assigned at birth
Enrollment: 46 (Actual)
Dates: Start 2024-01-28 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Improvements in Global longitudinal strain | at 8 weeks follow up
  GLS value was evaluated pre and post intervention. Pre intervention GLS were examined within the first 24 hour after PPCI, GLS post intervention at 8 weeks follow up GLS assesed with Epiq 7C ultrasound machine manufactured by Philips Medical Systems, the investigators conducted two-dimentional speckle-tracking investigations. These studies utilized QLAB/automated cardiac motion quantification (ACMQ) version 10.85 and QLAB/LV auto-strain version 12.0, both developed by Philips Healthcare. Three sequential cardiac cycles of apical 4, 2, and 3 chamber view images were stored using all scanners with the best machine settings and frame rates 50-70 frames per second for the purpose of measuring strain using speckle tracking echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Ilham Uddin, Medical Doctor, cardiologist, Principal Investigator — University of Diponegoro
Locations (1):
- Dr. Kariadi Central General Hospital, Semarang, Central Java, Indonesia

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT06661018/Prot_SAP_ICF_000.pdf